CLINICAL TRIAL: NCT06346210
Title: Optimal Timing for Tracheostomy in Invasively Mechanically Ventilated COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Healthcare Region Dalarna (Unknown)
Responsible Party: Sponsor
Other Study IDs: UNT: U1111-1288-2037
Record Dates: First submitted 2024-04-02; First posted 2024-04-03 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: COVID-19
Keywords: Critical care; Tracheostomy; Mechanical ventilation
MeSH Terms: conditions — COVID-19 | interventions — Tracheostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Not tracheostomised: Invasively mechanically ventilated COVID-19 patients who did not receive a tracheostomy within 60 days from tracheal intubation.
- Tracheostomised: Invasively mechanically ventilated COVID-19 patients who did receive a tracheostomy within 60 days from tracheal intubation.
  Interventions: Procedure: Tracheostomy

INTERVENTIONS:
Procedure: Tracheostomy — Surgery for tracheostomy
  Groups: Tracheostomised

SUMMARY:
Tracheostomy is a medical procedure performed on the front of a persons neck. It is used to create a connection between the persons trachea and a mechanical ventilator instead of using a tube going through the mouth into the trachea, oral intubation. Living with a tracheostomy tube is less stressful compared to oral intubation and facilitate being awake and the start of training on spontaneous ventilation in mechanically ventilated patients. Studies of the timing of tracheostomy are either severely affected by methodological bias of to small to determine an effect. Thus, it is not known what the optimal timing of the tracheostomy is in mechanically ventilated COVID-19 patients.

DETAILED DESCRIPTION:
Hypothesis It is hypothesised that timing of tracheostomy to day 9-11 is independently linked to a higher number of days, alive without invasive mechanical ventilation and several secondary outcomes when adequate methods to neutralize waiting time and immortal time bias are used.

Data sources Existing data provided for another project will be used.

Statistical methods:

A cohort study with a target trial emulation (1) on a dataset with cloned individuals assigned to different treatment strategies (i.e. tracheostomy at different timings). Censoring at deviation from assigned strategy or death (2). Adjustment for confounding will be used.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* admitted to an intensive care unit in Sweden from 2020 to 2021
* Main discharge diagnosis COVID-19 (ICD-10, U07.1)
* Invasive mechanical ventilation

Exclusion Criteria:

* No Swedish personal identification number.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Invasively mechanically ventilated adults in the Swedish intensive care registry.
Sampling Method: Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Ventilator free days alive | 60 days.
  Days alive without invasive mechanical ventilation during the first 60 days from start of invasive mechanical ventilation

SECONDARY OUTCOMES:
60 day mortality | 60 days.
  Mortality from any cause within 60 days from start of invasive mechanical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Björn Ahlström, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual patient data will be shared under the regulations of the European general data protection act and after researchers obtain relevant permissions from the Swedish ethical review authority.

REFERENCES:
- [Background] Hernan MA, Robins JM. Using Big Data to Emulate a Target Trial When a Randomized Trial Is Not Available. Am J Epidemiol. 2016 Apr 15;183(8):758-64. doi: 10.1093/aje/kwv254. Epub 2016 Mar 18. PMID 26994063
- [Background] Fu EL, Evans M, Carrero JJ, Putter H, Clase CM, Caskey FJ, Szymczak M, Torino C, Chesnaye NC, Jager KJ, Wanner C, Dekker FW, van Diepen M. Timing of dialysis initiation to reduce mortality and cardiovascular events in advanced chronic kidney disease: nationwide cohort study. BMJ. 2021 Nov 29;375:e066306. doi: 10.1136/bmj-2021-066306. PMID 34844936